CLINICAL TRIAL: NCT01734954
Title: Comparison of Two Techniques of Ultrasound-guided Sciatic Nerve Block Using Levobupivacaine 0.5% in Orthopedic Surgery at the Hospital Pablo Tobon Uribe - Clínica CES, 2013, Randomized Clinical Trial
Brief Title: Comparison of Two Techniques of Sciatic Nerve Block With Levobupivacaine 0.5% in Orthopedic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CES University (Other)
Collaborators: Hospital Pablo Tobón Uribe (Other); Clínica CES (Unknown)
Responsible Party: Principal Investigator, Marta Inés Berrío Valencia, Anesthesiologist, CES University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IACES
Record Dates: First submitted 2012-11-10; First posted 2012-11-28 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Anesthesia
Keywords: Nerve block; Sciatic nerve; Ultrasonography; Orthopedics; Hallux Valgus; Amputation; Arthrodesis; Arthroscopy; Fracture fixation; Osteotomy; Tendon transfer; Tenodesis; Tenotomy; Orthopedic procedure
MeSH Terms: conditions — Hallux Valgus; Ankylosis | interventions — Levobupivacaine; Anesthetics, Local; Ultrasonography; Oxygen; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sciatic nerve blockade at bifurcation (Experimental): Ultrasound-guided block at the bifurcation of the sciatic nerve
  Interventions: Procedure: Sciatic nerve anesthesia blockade at bifurcation.; Drug: Levobupivacaine 0.5%: 20 ml; Device: Portable Ultrasound Machine: Sonosite, M-Turbo, Bothell, WA; Device: Insulated Needle, (Stimuplex; Braun, Melsungen, Germany); Drug: supplemental oxygen; Drug: Midazolam; Drug: Intravenous analgesics; Procedure: Saphenous nerve block
- Sciatic block 2 cm beyond bifurcation (Experimental): Ultrasound-guided block of the sciatic nerve 2 cm beyond of the bifurcation
  Interventions: Procedure: Sciatic nerve blockade 2 cm beyond the bifurcation; Drug: Levobupivacaine 0.5%: 20 ml; Device: Portable Ultrasound Machine: Sonosite, M-Turbo, Bothell, WA; Device: Insulated Needle, (Stimuplex; Braun, Melsungen, Germany); Drug: supplemental oxygen; Drug: Midazolam; Drug: Intravenous analgesics; Procedure: Saphenous nerve block

INTERVENTIONS:
Procedure: Sciatic nerve anesthesia blockade at bifurcation. — A proximal and distal initial scan and define the site to block the bifurcation. A puncture with an insulated needle guided by ultrasound and injection of levobupivacaine circumferential in 0.5% and a total volume of 20 mL.
  Other Names: Sciatic Nerve Block
  Arms: Sciatic nerve blockade at bifurcation
Procedure: Sciatic nerve blockade 2 cm beyond the bifurcation — A proximal and distal initial scan and define the sites to block: tibial and peroneal nerves separate distal 2 cm from the bifurcation site. A puncture with an insulated needle guided by ultrasound and injection of levobupivacaine circumferential in 0.5% 10 mL tibial nerve and 10 mL to the peroneal nerve.
  Other Names: Sciatic nerve block
  Arms: Sciatic block 2 cm beyond bifurcation
Drug: Levobupivacaine 0.5%: 20 ml — Levobupivacaine is a local anesthetic that is commonly use for anesthesia nerve blockade.
  Other Names: Local Anesthetic
Device: Portable Ultrasound Machine: Sonosite, M-Turbo, Bothell, WA — An ultrasound machine is a device that is widely used for the correct placement of the local anesthetic for anesthesia nerve blockade.
  Other Names: Ultrasound
Device: Insulated Needle, (Stimuplex; Braun, Melsungen, Germany) — This is a specific kind of needle that is widely used for anesthesia nerve blockade.
  Other Names: Nerve blockade needle short bevel.
Drug: supplemental oxygen — supplemental oxygen during the block and/or during surgery
  Other Names: oxygen
Drug: Midazolam — Intravenous midazolam for sedation during the block and/or during surgery
Drug: Intravenous analgesics — Intraoperative administration intravenous of dipyrone 30-50 mg/Kg and or intravenous ketoprofen 100 mg or diclofenac 75 mg or ketorolac 30 mg
Procedure: Saphenous nerve block — Depending on sensitive territory committed by the type of surgery suprapatellar saphenous nerve block guided by ultrasound with 100 mm Stimuplex needle and injection of levobupivacaine 0.5% (total volume: 5 ml).

SUMMARY:
The purpose of this study is to evaluate the latency period (timing between the injection of the local anesthetic and the onset of complete sensory nerve block) of two approaches for ultrasound-guided popliteal sciatic nerve block: One of the approaches is the injection of the anesthetic just at the site of the bifurcation of the sciatic nerve and the other one is injecting the local anesthetic at least 2 cm beyond the bifurcation of the aforementioned nerve. Our main hypothesis is that the first approach will decrease the latency period, and probably, will increase the success rate of the nerve block as well as patient satisfaction.

DETAILED DESCRIPTION:
Compare the effectiveness of nerve blockade at the bifurcation site of the sciatic nerve versus distal (tibial and peroneal) using only levobupivacaine 0.5%. The primary outcome is the latency period of the nerve blockade; the secondary outcomes are rate of success of the procedure as well as patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ankle or foot surgery at Hospital Pablo Tobón Uribe and Clínica CES.
* Physical status classification of the American Society of Anesthesiologists (ASA) 1-3.
* Age: 18-70 years.
* Weight: 40-100 kg
* Taller than 140 cm.

Exclusion Criteria:

* No patient acceptance.
* Contraindications for nerve block (coagulopathy, local anesthetics allergy, sepsis, infection at the site of puncture).
* Neuropathy or myopathy affecting the lower limb.
* Psychiatric or neurological diseases that alter the evaluation of patient.
* Arrhythmias.
* Heart failure.
* Diabetes Mellitus.
* Pregnancy.
* Language barriers.
* Anticoagulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Latency period of sciatic nerve block. | 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes and 30 minutes after nerve block.
  Once the nerve blockade is done, a sensory evaluation will be performed in the surgical area every five minutes to determine the onset of the sensory nerve blockade in minutes.

SECONDARY OUTCOMES:
Success of sciatic nerve block | Every 5 minutes until 30 minutes until the end of the procedure for the nerve block; an additional measure will be performed at the end of of the surgery.
  The time to achieve a complete sensory nerve block, reached maximum at 30 minutes, in full distribution of tibial nerve and common fibular nerve for anesthesia.
Patient satisfaction | Postoperative 24 hours
  Using a categorical score we will measure satisfaction of nerve-block-procedure satisfaction and analgesia quality one day after surgery: patients will choose one of three options: no satisfied, satisfied or very satisfied.
Sensory block | 5, 10, 15, 20, 25 and 30 minutes after the block is finished
  Evaluation in 5, 10, 15, 20, 25 and 30 minutes after the procedure in the distribution of the common peroneal and tibial nerves
  0: Complete sensory block
  1. Almost complete sensory block: Decreased sensation to pinprick with a 24 gauge hypodermic needle
  2. Feeling normal (for each component: tibial and common peroneal) compared with the contralateral leg
Motor block | 5, 10, 15, 20, 25 and 30 minutes of completion after the block is finished
  Evaluation in 5, 10, 15, 20, 25 and 30 minutes after the procedure in the distribution of the common peroneal and tibial nerves 0: Complete motor blockade
  1. Motor block almost complete
  2. No motor block (for the tibial component for plantarflexion and dorsiflexion with the common peroneal) compared with the contralateral leg
First analgesic | 5 minutes, 30 minutes, 24 hours postoperative
  Time of first analgesic requirement in postoperative
Visual analog scale at rest | 5 minutes, 30 minutes, 24 hours postoperative
  Pain rating ranging from zero to ten VAS 0: no pain VAS 1-3: Mild pain VAS 4-6: Moderate Pain VAS 7-10: Severe pain
Dynamic visual analog scale | 5 minutes, 30 minutes, 24 hours postoperative
  Pain rating ranging from zero to ten with the movement
Intraneural injection | At the time of injection and execution of the block
  Increased diameter nerve or visualized by ultrasound visualization of the needle into the nerve at the time of injection
Vascular puncture | During the execution of the block
  Puncture of one or more blood vessels to visualize the needle within the vessel or to aspirate blood during block
Paresthesia during the procedure | At the time of the execution of the block
  Paresthesia during the procedure
Systemic toxicity of local anesthetics | During the execution of the block and 30 minutes after it
  Systemic toxicity of local anesthetics
Hematoma | During and inmmediately after the execution of the block
  Hematoma
Muscle weakness | 24 hours postoperative
  Subjective reduction in muscle strength at 24 hours postoperative
Altered sensitivity | 24 hours postoperative
  Subjective decreased sensitivity at 24 hours postoperative
Cramps postoperative | 24 hours postoperative of the block
  Feeling cramps within 24 hours of the block
Punctures | During the block
  Number of skin punctures during the block
Time for the execution of nerve block | In minutes: Time from placement of the transducer for the initial scan to final withdrawal of the needle
  Time from placement of the transducer for the initial scan to final withdrawal of the needle

CONTACTS AND LOCATIONS:
Overall Officials: Marta I Berrio, MD, Principal Investigator — CES University, Medellín, Antioquia, Colombia
Locations (2):
- Colombia (2):
  - Hospital Pablo Tobón Uribe, Medellín, Antioquia
  - Clínica CES, Medellín, Antioquia